CLINICAL TRIAL: NCT01727128
Title: A Phase I, Multicenter, Open-label, Single-dose, Parallel Group Study to Assess the Pharmacokinetics of BKM120 in Subjects With Mild, Moderate and Severe Hepatic Impairmen
Brief Title: Pharmacokinetic Study of BKM120 in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CBKM120C2104; 2011-002311-28 (EudraCT Number)
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2014-04

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; Clinical pharmacology study; Volunteer study
MeSH Terms: interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mild Hepatic Impaired Group (Experimental): Subjects can only be enroled into this group if they fit the Child -Pugh score criteria of severity category - mildly hepatically impaired
  Interventions: Drug: BKM120
- Moderate Hepatic Impaired group (Experimental): Subjects can only be enroled into this group if they fit the Child -Pugh score criteria of severity category - moderately hepatically impaired
  Interventions: Drug: BKM120
- Severe Hepatic Impaired Group (Experimental): Subjects can only be enroled into this group if they fit the Child -Pugh score criteria of severity category - Severely hepatically impaired
  Interventions: Drug: BKM120
- Control Group (Experimental): Matching healthy control subjects who do not have hepatic impairment and are matched to the hepatic impaired subjects by sex, age, gender and BMI
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120

SUMMARY:
To assess pharamcokinetics, safety and tolerability of a single oral dose of BKM120 in subjects with mild, moderate and severe hepatic impairment

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be in good health (except for additional/ specific inclusion criteria related to hepatic impaired subjects) as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests of no significance at screening
* Subjects must weigh at least 45 kg to participate in this study, and must have a body mass index (BMI) from (18.5-35.0 kg/m2)
* Subjects must be able to communicate well with the investigator, to understand the requirements of the study and agree to use strict contraception for 16 weeks after the last BKM120 dose

  ---Additional inclusion criteria Group 1 - control healthy subjects
* Subjects should be matched to the hepatic impaired subjects of group 2 in gender, age (± 10 years), weight (± 20%), and BMI (±5%)

  ---Additional inclusion criteria Group 2 - hepatic impaired subjects
* Subjects with physical signs consistent with stable hepatic impairment
* Child-Pugh Clinical Assessment Score consistent with degree of hepatic impairment (mild , moderate or severe)
* Subjects must be free of significant medical disorders unrelated to the subject's hepatic disorder as judged by the investigator.
* Absolute neutrophil count (ANC) ≥ 1.5 x 109 /L
* Platelet count ≥ 50 x 109 /L
* serum creatinine ≤ 1.5 x ULN

Exclusion Criteria:

* Significant illness, including infections, or hospitalization within the 2 weeks prior to dosing, except for the hepatic impaired subjects who due to their liver disease may be affected by significant medical problems which require frequent hospitalizations. Invasive systemic fungal infections need to be fully resolved prior to study entry
* Use of tobacco products within 2 weeks prior to dosing or during the study.
* Consumption of alcohol within 2 days prior to dosing or during the study
* Subjects with known ongoing alcohol and or/drug abuse within 1 month prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during screening and/or at baseline
* Subjects not willing to avoid certain study prohibited food, drink, over the counter medicines and supplements
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study.
* Medical history of cardiac disease and/or clinically significant ECG abnormalities.
* History of clinically significant hematologic, renal, endocrinologic, pulmonary cardiovascular, hepatic, or allergic disease medically documented
* Medical history of relevant psychiatric disorders
* Subjects with Diabetes Mellitus or subjects with glucose levels out of normal range as judge by the investigator
* History of immunodeficiency diseases, including Human Immunodeficiency Virus (HIV), as confirmed by (HIV-1, HIV-2) test

  * Additional exclusion criteria Group 1 (matched healthy control subjects) History or presence of liver disease or liver injury as indicated by an abnormal liver function profile A positive Hepatitis C test or a positive Hepatitis B surface antigen (HBsAg)
  * Additional exclusion criteria Group 2- hepatic impaired subjects
* Subjects with clinically significant abnormal findings, not consistent with clinical disease, upon physical examination, ECG or laboratory evaluation
* Any evidence of progressive liver disease (within the last 4 weeks prior to the screening visit) as indicated by liver transaminases, alkaline phosphatase and GGT or a ≥ 50% worsening of serum bilirubin or prothrombin time
* Total bilirubin > 6mg/dl
* Subject has ascites requiring intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of pharmacokinctis (PK) parameter Tmax | predose,0.5,1,1.5,2,3,4,6,8,12,24,48,72,96,144,192,240,288,336 hours post dose
  Measurment of effect of liver impairment on PK of BKM120 by assessment of the PK parameter TMax (time to maximum concentration)
Plasma concentration of PK parameter Cmax | predose,0.5,1,1.5,2,3,4,6,8,12,24,48,72,96,144,192,240,288,336 hours post dose
  Measurment of effect of liver impairment on PK of BKM120 by assessment of the PK parameter CMax (maximum concentration)
Plasma concentration of PK parameter AUC-t | predose,0.5,1,1.5,2,3,4,6,8,12,24,48,72,96,144,192,240,288,336 hours post dose
  Measurment of effect of liver impairment on PK of BKM120 by assessment of the PK parameter AUC-t (Area under the curve at specified timepoint) The specific key measure(s) or observation(s) that will be used to determine the effect of the intervention(s). Example: Change in left ventricular end systolic volume (LVESD) as measured by echocardiography Time to tumor progression Overall tumor response
Plasma concentration of PK parameter AUC-last | predose,0.5,1,1.5,2,3,4,6,8,12,24,48,72,96,144,192,240,288,336 hours post dose
  Measurment of effect of liver impairment on PK of BKM120 by assessment of the PK parameter AUC-last (Area under the curve at last timepoint) The specific key measure(s) or observation(s) that will be used to determine the effect of the intervention(s). Example: Change in left ventricular end systolic volume (LVESD) as measured by echocardiography Time to tumor progression Overall tumor response
Plasma concentration of PK parameter AUC-inf | predose,0.5,1,1.5,2,3,4,6,8,12,24,48,72,96,144,192,240,288,336 hours post dose
  Measurment of effect of liver impairment on PK of BKM120 by assessment of the PK parameter AUC-inf (Area under the curve to time infinity)
Plasma concentration of PK parameter CL/F | predose,0.5,1,1.5,2,3,4,6,8,12,24,48,72,96,144,192,240,288,336 hours post dose
  infMeasurment of effect of liver impairment on PK of BKM120 by assessment of the PK parameter CL/F (clearance)
Plasma concentration of PK parameter Vz/F | predose,0.5,1,1.5,2,3,4,6,8,12,24,48,72,96,144,192,240,288,336 hours post dose
  FMeasurment of effect of liver impairment on PK of BKM120 by assessment of the PK parameter Vz/F (Volume distribution)
Plasma concentration of PK parameter terminal T 1/2 | predose,0.5,1,1.5,2,3,4,6,8,12,24,48,72,96,144,192,240,288,336 hours post dose
  Measurment of effect of liver impairment on PK of BKM120 by assessment of the PK parameter terminal T 1/2 (terminal half-life)

SECONDARY OUTCOMES:
Adverse events severity | From baseline day-1 to 30 days post dose
  Severtiy of adverse events severity based on the CTCAE criteria to assess safety and tolerability of a single dose of BKM120
Change from baseline in laboratory parameters | From baseline day-1 to 30 days post dose
  Change from baseline in hematological and biochemical laboratory parameters
Change from baseline in ECG parameters | From baseline day-1 to 30 days post dose
  Change from baseline in ECG parameters
Change from baseline between PK parameters and total bilirubin, prothrombin time or INR and serum albumin | From baseline day-1 to 15 days post dose
  Relationship between PK parameters and baseline hepatic function parameters
measurement of plasma binding | From baseline day-1 to 15 days post dose
  Determination of the free fraction of BKM120 in plasmaexpressed weher relevant in terms of unbound drug concentration
Adverse events frequency | From baseline day-1 to 30 days post dose
  Frequency of adverse events severity based on the CTCAE criteria to assess safety and tolerability of a single dose of BKM120

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Moscow, Russia

REFERENCES:
- See also: Results for CBKM120C2104 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12183